CLINICAL TRIAL: NCT00639873
Title: Artemisinin Resistance in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); World Health Organization (Other)
Responsible Party: Principal Investigator, Harald Noedl, Assoc. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUW # 83/2008
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Malaria
Keywords: Uncomplicated P. falciparum malaria
MeSH Terms: conditions — Malaria | interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AS 2mg/kg (Experimental): Artesunate monotherapy 2mg/kg/day for 7 days
  Interventions: Drug: Artesunate
- AS 4mg/kg (Experimental): Artesunate monotherapy 4mg/kg/day for 7 days
  Interventions: Drug: Artesunate
- QD Control (Active Comparator): Quinine-doxycycline for 7 days
  Interventions: Drug: quinine-doxycycline

INTERVENTIONS:
Drug: Artesunate — 2 or 4 mg/kg/day for 7 days
  Arms: AS 2mg/kg; AS 4mg/kg
Drug: quinine-doxycycline — quinine-doxycycline for 7 days
  Arms: QD Control

SUMMARY:
A randomized, controlled clinical trial conducted in Southeastern Bangladesh using artesunate monotherapy to determine the baseline sensitivity of P. falciparum to artemisinins.

DETAILED DESCRIPTION:
A total number of 100 volunteers with acute uncomplicated falciparum malaria will be randomly assigned one of 3 arms to be treated with artesunate monotherapy or quinine/doxycycline for 7 days at a ratio of 2:2:1. The study design will be based on the WHO recommendations for the 'Assessment and Monitoring of Antimalarial Drug Efficacy for the Treatment of Uncomplicated Falciparum Malaria' (WHO, 2003). Study participants will be otherwise healthy malaria patients aged 8 to 65 years with uncomplicated falciparum malaria recruited at the Bandarban Sadar Hospital, Bangladesh.

The artesunate will be administered orally (a single dose of 2 or 4 mg/kg/day) over a total duration of 7 days by directly observed therapy.

Patients will be admitted to the hospital for the duration of study drug administration or until all signs and symptoms of malaria have disappeared, whichever comes later. Thereafter they will be followed as outpatients until Day 42 with scheduled follow-up visits on Day 14, 28, 35, and 42.

In vitro drug sensitivity assays will be performed from samples on inclusion and in case of recrudescence. Drug levels will be measured on the first and last day of therapy.

Primary clinical outcome is cure (Adequate Clinical and Parasitological Response - ACPR) on Day 28 and 42. Secondary outcome measures are time until parasite, fever, and gametocyte clearance (PCT, FCT, and GCT). Parasite genotyping will be used to distinguish recrudescences from reinfections by PCR for patients in whom recrudescences cannot be fully excluded. Subjects will be monitored for clinical adverse events throughout the study duration.

Blood will be drawn on the day of admission (before initiating therapy) for in vitro drug sensitivity testing and for PCR (markers of drug resistance and to distinguish recrudescence from reinfection by genotyping). Malaria smears will be prepared twice daily until parasite clearance and on Days 7, 14, 21, 28, 35, and 42 or whenever symptoms consistent with malaria appear. Plasma samples for determining drug levels will be obtained on the first and last day of therapy. Study participation for each individual will be 42 days.

ELIGIBILITY:
Inclusion Criteria:

1. Acute symptomatic falciparum malaria infection as determined by malaria smear with a parasite density of 1,000 to 100,000 asexual parasites/uL as determined on the screening smear with fever (defined as ≥37.5C), or reported history of fever within the last 48 hours.
2. Age: 8-65 years old
3. All females between the age of 12 and 50 are required to have a negative human chorionic gonadotropin (hCG) pregnancy test (urine). All females of childbearing potential (not surgically sterile, or less than two years menopausal) are required to use an acceptable method of contraception throughout the study
4. Written informed consent obtained
5. Willing to stay under close medical supervision for the study duration of 42 days
6. Otherwise healthy outpatients

Exclusion Criteria:

1. Pregnant women, nursing mothers, or women of childbearing potential who do not use an acceptable method of contraception
2. Mixed malaria infection on admission by malaria smear
3. A previous history of intolerance or hypersensitivity to the study drugs or to drugs with similar chemical structures
4. Malaria drug therapy administered in the past 30 days by history
5. History of significant cardiovascular, liver or renal functional abnormality or any other clinically significant illness, which in the opinion of the investigator would place them at increased risk.
6. Symptoms of severe vomiting (no food or inability to take food during the previous 8 hours).
7. Signs or symptoms of severe malaria (as defined by WHO 2000)
8. Unable and/or unlikely to comprehend and/or follow the protocol

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Cure | 42 days
  Cure is defined as adequate clinical and parasitological response (ACPR) as opposed to early treatment failure / late treatment failure

SECONDARY OUTCOMES:
Treatment response | 42 Days
  Treatment response parameters: parasite, fever, and gametocyte clearance

CONTACTS AND LOCATIONS:
Overall Officials: Harald Noedl, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Bandarban Sadar Hospital, Bandarban Sadar, Bandarban, Bangladesh

REFERENCES:
- [Derived] Starzengruber P, Swoboda P, Fuehrer HP, Khan WA, Hofecker V, Siedl A, Fally M, Graf O, Teja-Isavadharm P, Haque R, Ringwald P, Noedl H. Current status of artemisinin-resistant falciparum malaria in South Asia: a randomized controlled artesunate monotherapy trial in Bangladesh. PLoS One. 2012;7(12):e52236. doi: 10.1371/journal.pone.0052236. Epub 2012 Dec 18. PMID 23272227
- See also: MARIB - Malaria Research Initiative Bandarban — http://www.marib.org
- See also: Medical University of Vienna — http://www.meduniwien.ac.at
- See also: ICDDR,B — http://www.icddrb.org